CLINICAL TRIAL: NCT05512845
Title: The Double Factor Technique: a Computer-guided Implant Surgery Technique for Fully Edentulous Patients
Acronym: DoubleFactor
Status: Completed | Type: Observational
Sponsor: Adrià Jorba García (Other)
Responsible Party: Sponsor-Investigator, Adrià Jorba García, Principal Investigator, University of Barcelona
Organization: University of Barcelona (Other)
Other Study IDs: Double Factor
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Surgery, Computer-Assisted; Dental Implants
Keywords: Dental Implants; Surgery, Computer-Assisted; Fully edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Double factor group: Patients treated with full arch implant supported prostheses based on the All-on-four® concept. All implants were placed using the "double factor" computer assisted surgery technique, which involves combination of the static and dynamic computer assisted surgery protocols.
  Interventions: Procedure: Double Factor technique

INTERVENTIONS:
Procedure: Double Factor technique — The "double factor" computer assisted surgery technique, involves the combination of the static and dynamic computer assisted surgery protocols to place dental implants in the same surgery.
  Other Names: Dynamic and static computer assisted surgery

SUMMARY:
To overcome the limitations of the current dynamic and static Computer Assisted surgery protocols in fully edentulous patients, and combine the advantages of both approaches, a new technique has been developed, referred to as the "double factor" technique.

This study consists in a single arm observational prospective clinical study and the aim was to assess the accuracy and patient's perception and quality of life of the "double factor" technique in treating fully edentulous patients.

DETAILED DESCRIPTION:
This is a prospective observational clinical study. Each patient enrolled in this study will be treated using the "all on four concept" using the double factor technique.

Preoperative virtual planification of dental implants on a pre-acquired cone beam computed tomography (CBCT) will be performed for each patient using the same system.

During the surgical phase, four dental implant will be placed in a fully guided approach using "the double factor technique. This technique merges the static and dynamic computer-guided surgical approach in the same surgery.

Then after the surgical procedure a PROMs questionnaire will be asked to the patients.

Finally, a postoperative CBCT will be performed and overlapped with the preoperative CBCT (with the implants planification) and implant position deviations between the planned and final position will be measured.

The study devices are CE- (Conformité Européenne, meaning European Conformity) marked products and used within their intended use.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous patients or with terminal dentition that requires an implant supported rehabilitation
* Healthy patients ASA I and II (American Society of Anesthesiologists classification)
* Over 18 years old patients

Exclusion Criteria:

* Partially edentulous patients
* Systemic or local conditions that contraindicates dental implant surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive edentulous patients or with terminal dentition treated with full arch implant supported prostheses based on the All-on-four® concept and the computer assisted surgery "double factor" technique will be included in the trial.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Angular deviation | The day of the surgery
  Angular deviation between the virtual planed position of the implant and the final implant position. Measured in degrees
Platform 3D deviation | The day of the surgery
  global deviation at the platform of the dental implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).
APex 3D deviation | The day of the surgery
  global deviation at the apex of the dental implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).
Platform 2D deviation | The day of the surgery
  Lateral deviation at the platform of the dental implant between the virtual planned position and the final position of the dental implant measured in 2 axes of the space (x and y, 2D deviation). Measured in millimeters (mm).
Apex depth deviation | The day of the surgery
  Depth deviation of the apex of the dental implant between the virtual planned position and the final position of the dental implant in the Z-axis. Measured in millimeters (mm).

SECONDARY OUTCOMES:
Patient-reported outcome measures (PROMs). | Seven postoperative days.
  Patients perception of their functional well-being and health status during the dental implant treatment with a the "double factor" technique. We will use OHIP-14 (Oral Health Impact Profile) questionnaire.
Patient-reported outcome measures (PROMs). | Seven postoperative days.
  Patients perception during the surgery will be assessed using a designed questionnaire (Likert scale)
Postoperative pain | Seven postoperative days.
  A registration of the postoperative pain using a Visual Analog Scale (VAS) from 0mm to 100mm, meaning 0mm no pain and 100mm the maximum pain.
Analgesic medication consumption record | Seven postoperative days.
  The patient will be asked to record all the analgesic medication intake during the first 7 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Adrià Jorba-García, DDS, MS, Principal Investigator — University of Barcelona; Carmen Pomares-Puig, MD, DDS, Study Chair — University of Valencia; M Angeles Sánchez-Garcés, MD, MS, PhD, Study Chair — University of Barcelona
Locations (1):
- Clinica Perio&Implant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vercruyssen M, Fortin T, Widmann G, Jacobs R, Quirynen M. Different techniques of static/dynamic guided implant surgery: modalities and indications. Periodontol 2000. 2014 Oct;66(1):214-27. doi: 10.1111/prd.12056. PMID 25123770
- [Background] Pomares-Puig C, Sanchez-Garces MA, Jorba-Garcia A. Dynamic and static computer-guided surgery using the double-factor technique for completely edentulous patients: A dental technique. J Prosthet Dent. 2022 Nov;128(5):852-857. doi: 10.1016/j.prosdent.2021.02.022. Epub 2021 Mar 31. PMID 33810850
- [Background] Pomares C. A retrospective study of edentulous patients rehabilitated according to the 'all-on-four' or the 'all-on-six' immediate function concept using flapless computer-guided implant surgery. Eur J Oral Implantol. 2010 Summer;3(2):155-63. PMID 20623040
- [Background] Jorba-Garcia A, Gonzalez-Barnadas A, Camps-Font O, Figueiredo R, Valmaseda-Castellon E. Accuracy assessment of dynamic computer-aided implant placement: a systematic review and meta-analysis. Clin Oral Investig. 2021 May;25(5):2479-2494. doi: 10.1007/s00784-021-03833-8. Epub 2021 Feb 26. PMID 33635397